CLINICAL TRIAL: NCT02730793
Title: Aztreonam Aerosol to Treat Cystic Fibrosis Nasal Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated due to an inability to recruit study subjects
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eastern Virginia Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM20005657
Record Dates: First submitted 2015-11-03; First posted 2016-04-06 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; P. aeruginosa (PA)
MeSH Terms: conditions — Cystic Fibrosis | interventions — Aztreonam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Therapy (Active Comparator): Oral Inhalation via PARI Altera Device: Standard Therapy Comparator (Oral Aztreonam 75mg three times a day) AND Nasal Inhalation via PARI PAS Device: Nasal Placebo-Normal Saline twice per day
  Interventions: Drug: Oral Aztreonam; Drug: Nasal Placebo
- Study Therapy (Experimental): Oral Inhalation via PARI Altera Device: Standard Therapy Comparator (Oral Aztreonam 75mg three times a day) AND Nasal Inhalation via PARI PAS Device: Experimental- Nasal Aztreonam 75 mg twice per day
  Interventions: Drug: Oral Aztreonam; Drug: Nasal Aztreonam

INTERVENTIONS:
Drug: Oral Aztreonam — Standard Therapy Comparator (Oral Cayston 75mg three times a day)
  Other Names: Cayston; Azactam
Drug: Nasal Aztreonam — Study Therapy (nasal Aztreonam 75mg twice per day)
  Other Names: Cayston; Azactam
  Arms: Study Therapy
Drug: Nasal Placebo — Placebo (nasal saline twice per day)
  Other Names: Saline
  Arms: Standard Therapy

SUMMARY:
This study is designed as a masked, two center, randomized, placebo-controlled pilot study to evaluate the safety and efficacy of nasal and oral inhalation of 75 mg aztreonam in subjects with CF and lung infection due to PA. The study will involve two sites: Virginia Commonwealth University Medical Center (VCU) and Eastern Virginia Medical School (EVMS). Potential subjects will be identified in each site's CF clinic.

DETAILED DESCRIPTION:
This study is designed to explore the efficacy and safety of nasal aztreonam administered using the Pari Sinus Nebulizer combined with oral Cayston aerosol therapy compared to placebo on clinical and laboratory endpoints such as risk of antibiotic-resistant Pseudomonas aeruginosa (PA), time to pulmonary infection exacerbation, nasal quality of life, pulmonary function, nasal and lower airway cultures, and properties of mucus.

P. aeruginosa (PA) is a primary cause of lung infections in persons with cystic fibrosis (CF) (1). Over the past decade, studies have shown that aerosolized antibiotics can reduce lower respiratory bacterial load, decrease exacerbations of pulmonary disease, and in many patients improve pulmonary function. Cayston (aztreonam) oral aerosol using the PARI Altera Nebulizer System was approved by the FDA in February 2010 for CF patients 7 years of age or older with PA (2). In 2011, 35.8% or patients in the National CF Patient Registry used Cayston for treatment (3). Bacterial cultures suggest that the upper airways and lower airways of CF patients are cross-infected by PA and that the paranasal sinuses can act as a bacterial reservoir (4). There is improved post-transplanation patient survival for recipients that undergo sinus surgery and daily nasal washes to reduce bacterial load (2).

Routine CF care does not generally include upper airway assessment. There are no published studies evaluating the effect of aerosol antibiotics to treat nasal and sinus infections in CF in combination with oral inhaled aerosol therapy to treat the lower airway disease. However Mainz and colleagues published a case report that suggested that sinonasal administration of tobramycin using the Pari Sinus nebulizer (Pari Corp, Starnberg, Germany) delayed PA lower respiratory infection in a 12 year-old with CF who had chronic mucopurulent rhinosinusitis (5) and studies in chronic obstructive pulmonary disease suggest that treating upper airways can also improve coexistent lower airway disease.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 7 years of age or older and able to perform pulmonary function testing
2. Confirmed diagnosis of CF by the 1997 CF Consensus Conference criteria and followed by the VCU or EVMS CF clinic
3. Presence of PA in 2 lower respiratory tract (sputum) cultures in the 24 months before screening
4. Subjects and/or parent guardian must be able to give written informed consent prior to any study related procedure
5. All sexually active female subjects who are of childbearing potential must agree to use an effective method of contraception (i.e.condoms or abstinence).
6. All sexually active female subjects must have a negative pregnancy test at screening (V0).
7. Clinically stable determined by the study physician with no significant new respiratory symptoms.
8. Presence of PA in nasal culture (swab or secretion) or sinus culture obtained in the 12 months before screening or at screening visit

Exclusion Criteria:

1. Use of oral, IV or inhaled antibiotics within 0 days before study other than low dose azithromycin
2. Severe pulmonary disease with FEV1<30% predicted of baseline SpO2<0.90
3. ENT surgery within 6 months of screening
4. Allergy or documented adverse reaction to aztreonam
5. Epistaxis or significant (>30mL) hemoptysis in the past 6 months
6. Frequent (weekly or more frequently) or severe headaches
7. Subject is unlikely to comply with the procedures scheduled in the protocol
8. Subject participates in another clinical trial within 30 days prior to study entry
9. Subjects who have had a lung transplant will be excluded
10. Prisoners will be excluded
11. Non-English Speaking patients will be excluded

Ages: 7 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce K Rubin, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Children's Hospital of Richmond at VCU, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be deidentified and will not be availalble.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Therapy | Study Therapy
Started | 2 | 3
Completed | 2 | 1
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Because of the low number of enrollees with only 1 in the treatment group, results are not reported to protect the confidentiality of the participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Therapy | Study Therapy | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Number of Protocol-defined Pulmonary Exacerbations Treated With IV Anti-pseudomonal Antibiotics on Day 140
Description: Protocol-Defined Pulmonary Exacerbation includes events that are characterized by change or worsening pulmonary symptoms (increased cough, increased sputum production and chest congestion, decreased appetite and exercise tolerance), loss of weight, and lung function decline that prompt initation of antibiotic therapy. Protocol-defined exacerbations in subjects that warrant treatment with IV antibiotics will be determined from the medical record during the course of this study.
Time Frame: 140 days
Population: as for baseline characteristics
Arm/Group | Standard Therapy | Study Therapy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time to First Protocol-defined Pulmonary Exacerbation Treated With IV Anti-pseudomonal Antibiotics
Description: Protocol-Defined Pulmonary Exacerbation includes events that are characterized by change or worsening pulmonary symptoms (increased cough, increased sputum production and chest congestion, decreased appetite and exercise tolerance), loss of weight, and lung function decline that prompt initation of antibiotic therapy. Protocol-defined exacerbations in subjects that warrant treatment with IV antibiotics will be determined from the medical record during the course of this study. The time of beginning the study to first protocol-defined pulmonary exacerbation will also be determined from the medical record during the course of this study.
Time Frame: Up to 6 months
Population: as for baseline characteristics
Arm/Group | Standard Therapy | Study Therapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Sinus and Nasal QoL Questionnaire (SNOT-20) on Day 140 and Day 168
Description: The Sino-Nasal Outcome Test 20 (SNOT-20) is a validated health-related QOL questionnarie designed to determine the impact of sinonasal dysfunction. Patients will assess nasal symptoms, emotion, and activity on a scale of worsening symptoms scored 1 through 7 to provide a quantifiable score capable of disease severity. It has been shown as a responsive measure of health-related quality of life and suitable for use in outcomes studies and routine clinical care. Survey responses from Day 140 and Day 168 will be compared to the SNOT20 survey responses from previous visits (V1, V2, and V4)
Time Frame: Day 140 and Day 168
Population: as for baseline characteristics
Arm/Group | Standard Therapy | Study Therapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Cystic Fibrosis QoL Score (CFQ-R) on Day 140
Description: The CFQ-R is a validated patient-reported outcome measuring health-related quality of life for children and adults with CF. The CFQ-R contains both general and CF-specific scales. The CFQ-R was administered at Visits 1, 6, and 7. The endpoint was change in CFQR on day 140 compared to V1 and V5.
Time Frame: Day 140
Population: as for baseline characteristics
Arm/Group | Standard Therapy | Study Therapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Pulmonary Function (FVC and FEV1 Percent Predicted) on Day 140
Description: Routine spirometry will be performed according to American Thoracic Society (ATS) guidelines. A minimum of three maneuvers will be performed. The largest FVC and FEV1 will be reported after examining data from all acceptable curves even if they did not originate from the same maneuver. Data will be expressed both in absolute values and as percent (%) predicted based upon NHANES predicted values.
Time Frame: Day 140
Population: as for baseline characteristics
Arm/Group | Standard Therapy | Study Therapy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Paired Sputum Cultures and Nasal Swabs for Bacteria and Antibiotic Resistance
Description: Expectorated sputum and nasal swabs will be cultured at each visit using standardized procedures to identify CF pathogens as well as susceptibility to a standard panel of antibiotics.
Time Frame: 1 year
Population: as for baseline characteristics
Arm/Group | Standard Therapy | Study Therapy
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Acoustic Rhinometry for Nasal Obstruction (Volume) (Will be Measured at VCU Site ).
Description: Acoustic rhinometry is used to measure cross-sectional volume of the nasal cavity allowing the calculation of nasal volume. Reflected sound waves are painlessly introduced through nasal adaptors into the nasal passages allowing the production of area-distance graphs.
Time Frame: 1 year
Population: as for baseline characteristics
Arm/Group | Standard Therapy | Study Therapy
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Safety and Adverse Events Including Nasal Stuffiness, Epistaxis, and Headache.
Description: The frequency, severity and duration of all nasal and pulmonary adverse events, regardless of cause, will be recorded in REDCap as an electronic case report form. Serious adverse events will be captured in OnCore. The frequency and severity of adverse events will be calculated for each patient, with each patient counted once using the most severe grade experienced. The duration of adverse events will be calculated by the number of days each event persisted. Tables will be generated for all adverse events including serious adverse events and withdraws from the study.
Time Frame: 1 year
Population: as for baseline characteristics
Arm/Group | Standard Therapy | Study Therapy
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Protocol-defined Pulmonary Exacerbations Treated With Oral Anti-pseudomonal Antibiotics
Description: Protocol-Defined Pulmonary Exacerbation includes events that are characterized by change or worsening pulmonary symptoms (increased cough, increased sputum production and chest congestion, decreased appetite and exercise tolerance), loss of weight, and lung function decline that prompt initation of antibiotic therapy. Protocol-defined exacerbations in subjects that warrant treatment with oral antibiotics will be determined from the medical record during the course of this study.
Time Frame: 1 year
Population: as for baseline characteristics
Arm/Group | Standard Therapy | Study Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Standard Therapy | Study Therapy
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT02730793/Prot_SAP_000.pdf